CLINICAL TRIAL: NCT01871129
Title: The Effects of Postoperative Dexmedetomidine Sedation to Haemodynamics During Extubation
Brief Title: The Effects of Dexmedetomidine to Postoperative Awakening and Extubation-related Changes in Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R13046M
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Dexmedetomidine; Postoperative Period; Airway extubation; Systolic Pressure
MeSH Terms: conditions — Hypertension | interventions — Dexmedetomidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline group (Placebo Comparator): Difference from the normal protocol actualizes at the point when propofol infusion is cut off. From there on the patient in this group receives saline infusion up to the point where 15 minutes have passed after the extubation procedure.
  Interventions: Other: Saline (placebo)
- Dexmedetomidine group (Active Comparator): Difference from the normal protocol happens when normally the propofol infusion is cut off. From there on the patient in this group receives dexmedetomidine infusion up to the point where 15 minutes have passed after the extubation procedure.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be diluted into a saline solution to a recommended concentration of 4 micrograms per millilitre. The saline will then be initially administered at the rate of 0.5 micrograms/kg/h and from that point the amount will be reduced to the point where the patient breathes well and is calm (compare dexmedetomidine recommendation at 0.2-1.4 ug/kg/h). The infusion rate will then be approximately 1-10 ml/h for a patient of 80 kgs weight. The exact dosage cannot be predetermined because it differs in each individual. In the control group the infusion speed is matching.
  Other Names: Dexdor
  Arms: Dexmedetomidine group
Other: Saline (placebo) — Saline placebo infusion will be adjusted the same fashion as the active comparator drug.
  Other Names: Saline 0,9%; Normal saline
  Arms: Saline group

SUMMARY:
The postoperative removal of intubation tube induces a noticeable sympathic response and increase of blood pressure. The risk of complications is especially elevated with the patients having cardiac surgery. Though sedation inhibits the sympathetic responses to extubation, according to the current protocol the propofol infusion has to be discontinued well before extubation because of its inhibitory effects on breathing centers.

Dexmedetomidine is relatively new anesthesia drug. Dexmedetomidine is unique in its characteristic that it does not have the paralyzing effect on breathing. The aim of our study is to work out whether dexmedetomidine-extended propofol sedation over the extubation diminishes the aforementioned harmful effects of the extubation procedure.

Study design is prospective double-blinded randomized study. The investigators compare two groups of 25 patients (total 50), who are of 60-90 years of age and are having either aortic valve surgery or the mentioned accompanied with cardiopulmonary bypass operation. The first group receives dexmedetomidine infusion and the other receives placebo infusion after the end of propofol infusion.

The specific goal of the study is to figure what haemodynamic - mostly blood pressure related - changes can be observed when the postoperatively cut propofol infusion is continued with dexmedetomidine over the extubation procedure.

Our hypothesis is that by using dexmedetomidine supplemented sedation the normally notifiable peak in blood pressure may be avoided.

The study will be carried out completely in Cardiac ICU in Tampere University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient has to be scheduled for aortic valve surgery OR previous AND coronary artery bypass
* Patient has to be 60 to 90 years of age

Exclusion Criteria:

* If a patient is unable to give informed concent to participate the study
* If a patient is allergic or otherwise hypersensitive to the drug used in the study
* If the patient has either insufficient kidney or insufficient liver function

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Highest value of systolic blood pressure during extubation period | Starting five minutes before the extubation, lasting up to 1.5 hours.
  The values of this variable will be collected from the point when propofol infusion is cut. This data will be used to estimate the base level of SAP for further analysis within this study.

SECONDARY OUTCOMES:
Risk index calculated from systolic blood pressure value and time spent in that value. | Starting at the point when propofol infusion is halted and lasting up to three hours after extubation.
  With the risk index we are better able to assess the total risk of the high levels of blood pressure to the patient. The risk index is dependant on the time integral of the blood pressure, for which the zero-value may be calculated from average pre-extubation SAP level.

CONTACTS AND LOCATIONS:
Overall Officials: Kati M Järvelä, MD PhD, Principal Investigator — TAYS Sydänkeskus Oy (Heart Center CO. Tampere University Hospital)
Locations (1):
- TAYS Sydänkeskus Oy (Heart Center CO. Tampere University Hospital), Tampere, Finland